CLINICAL TRIAL: NCT04698343
Title: Exploratory Study Assessing the Response of Restless Legs Syndrome (RLS) Patients to Non-invasive Peripheral Nerve Stimulation (NPNS) During Opioid Medication Reduction
Brief Title: Noninvasive Peripheral Nerve Stimulation for Restless Legs Syndrome During Opioid Medication Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noctrix Health, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-03; R44NS117294 (NIH)
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Noninvasive Peripheral Nerve Stimulation (NPNS) (Experimental): NPNS device programmed to deliver active stimulation.
  Interventions: Device: Noninvasive Peripheral Nerve Stimulation (NPNS)

INTERVENTIONS:
Device: Noninvasive Peripheral Nerve Stimulation (NPNS) — NPNS device programmed to deliver active stimulation.

SUMMARY:
Prospective open-label single-arm feasibility study assessing the tolerability of opioid medication reduction in conjunction with noninvasive peripheral nerve stimulation (NPNS) for patients taking prescription opioids to treat moderate-severe primary RLS.

DETAILED DESCRIPTION:
For RLS patients taking a stable dose of prescription opioid medications prior to study entry, iterative opioid dose reduction is performed in conjunction with open-label NPNS treatment. For each of two iterative step-downs in opioid dose (step-down #1 and step-down #2), a 1-2-week run-in phase to allow resolution of opioid withdrawal symptoms unrelated to RLS is followed by a 1-wk assessment phase to evaluate if RLS symptoms have increased. Study participation is terminated if there is a clinically significant increase in RLS severity during the assessment phase or if there are intolerable opioid withdrawal symptoms at any time. Participants who tolerate both step-downs have the option of an extension phase involving a third step-down with the same format.

ELIGIBILITY:
Inclusion Criteria:

* Subject has received a medical diagnosis of primary restless legs syndrome (RLS)
* Subject is currently taking a stable dose of at least one prescription opioid for RLS, where the total opioid dose is less than or equal to 60mg morphine milligram equivalents (MME) per day.
* RLS symptoms are most significant in the subject's legs and/or feet.
* Subject possesses the necessary equipment, internet/phone accessibility, and communication ability to complete electronic questionnaires and respond to electronic communications and phone calls from the research staff throughout the in-home portion of the study.
* Subject is 18 to 89 years of age (inclusive) when written informed consent is obtained.
* Subject has signed a valid, Institutional Review Board (IRB)-approved informed consent form, can understand the requirements of the study and instructions for device usage, and can converse in English.
* Subject has been taking a stable dose and schedule of prescription opioids for RLS for at least 3 months prior to enrollment.

Exclusion Criteria:

* Subject has RLS that is known to be caused by another diagnosed condition (i.e. secondary RLS).
* Subject was misdiagnosed with RLS, as determined by the investigator (e.g. actual diagnosis of Periodic Leg Movement Disorder (PLMD), arthritis, leg spasms or neuropathy without comorbid RLS).
* Subject has primary sleep disorder other than RLS that significantly interferes with sleep at the present time (e.g. unmanaged sleep apnea or general insomnia).
* Subject has been diagnosed with one of the following conditions at any time: Epilepsy or other seizure disorder, Severe movement disorder symptoms (Parkinson's disease, Huntington's disease, dyskinesia, dystonia), Deep Vein Thrombosis, Multiple sclerosis
* Subject has an active diagnosis of one of the following conditions: Acute or chronic infection other than viral upper respiratory tract infections, Stage 4-5 chronic kidney disease or renal failure, Iron-deficient anemia, Severe edema affecting lower legs
* Subject has any of the following at the location of device application: Acute injury, Cellulitis, Open sores
* Subject has a malignancy within the past 5 years (not including basal or squamous cell skin cancer)
* Subject is on dialysis or anticipated to start dialysis while participating in the study
* Subject has severe peripheral neuropathy affecting the lower legs and/or subject has neuropathy and is unable to clearly distinguish between symptoms of neuropathy and symptoms of RLS.
* During NPNS calibration, subject has a sensation threshold above the upper-cutoff value (e.g. 30mA), the subject finds stimulation intensities less than 15 mA to be uncomfortable or distracting, or the device does not properly fit the subject.
* Subject has significantly changed dose or schedule of a medication that may impact RLS symptoms within the 30 days prior to enrollment, as judged by the investigator (e.g. antidepressants, sleep medications, sedative antihistamines).
* Subject has received an investigational drug or device within the last 30 days or is planning to receive an investigational device during the duration of the study.
* Subject has another medical condition that may affect validity of the study as determined by the investigator.
* Subject is unable or unwilling to comply with study requirements.
* Moderate or severe cognitive disorder or mental illness.
* Subject has prior experience with Noctrix Health NPNS devices.
* Subject has active implantable medical devices anywhere in the body (including pacemakers), or metal implant at the site of study device electrode application.
* Subject has known allergy to electrode gel, polyurethane foam, or lycra.
* Subject is pregnant or trying to become pregnant.
* Subject has undergone a major surgery (excluding dental work) in the previous 30 days.
* Subject has another medical condition that may put the subject at risk as determined by the investigator.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Charlesworth, PhD, Study Director — Noctrix Health, Inc.
Locations (2):
- United States (2):
  - Mark J Buchfuhrer private practice, Downey, California
  - Ohio Sleep Medicine Institute, Dublin, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchfuhrer MJ, Roy A, Rodriguez S, Charlesworth JD. Adjunctive tonic motor activation enables opioid reduction for refractory restless legs syndrome: a prospective, open-label, single-arm clinical trial. BMC Neurol. 2023 Nov 21;23(1):415. doi: 10.1186/s12883-023-03462-6. PMID 37990163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20-40 planned, 21 enrolled, 20 analyzed
  [1 enrolled in planned pilot phase, not part of analysis]
Pre-assignment Details: Participants undergo an iterative opioid dose reduction alongside open-label NPNS administration. Each of the two dose step-downs (Phase 1 and Phase 2) involves a 1-2-wk run-in period followed by a 1-wk assessment. This ensures resolution of opioid withdrawal symptoms and confirms NPNS usage instructions. Study ends if RLS severity increases or not tolerated. Those tolerating both phases may opt for a third dose reduction extension.
Period: Overall Study
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Started | 20
Completed Phase 1 | 14
Completed Phase 2 | 4
Completed Phase 3 | 3
Completed | 3
Not Completed | 17
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 2
Not completed — Failed to meet the required reduction in opioid dosage due to increased RLS symptoms | 4
Not completed — 1 was discontinued based on CGI-I score exceeding 5 | 1
Not completed — Personal reasons | 3
Not completed — 1 withdrew due to non-RLS opioid withdrawal symptoms | 1

BASELINE CHARACTERISTICS:
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
IRLS total score at baseline, mean (SD) [Mean (Standard Deviation); unit: units on a scale] | 9.8 (8.5)
Duration of RLS symptoms, mean (SD), y [Mean (Standard Deviation); unit: years] | 31.1 (14.1)
Number of prior RLS medications, mean (SD) [Mean (Standard Deviation); unit: number of RLS medications] | 3.2 (1.6)
Prior RLS medications, n (%) - Dopamine agonist [Count of Participants; unit: Participants] | 19
Prior RLS medications, n (%) - Alpha-2-delta ligand [Count of Participants; unit: Participants] | 12
Prior RLS medications, n (%) - Benzodiazepine [Count of Participants; unit: Participants] | 4
Prior RLS medications, n (%) - Opioid [Count of Participants; unit: Participants] | 2
Duration of opioid treatment for RLS, mean (SD), years [Mean (Standard Deviation); unit: years] | 8.0 (4.6)
Baseline opioid dosage, mean (SD), Morphine Milligram Equivalents (MME) [Mean (Standard Deviation); unit: MME] | 39.0 (15.6)
Current RLS medications, n (%) - Methadone [Count of Participants; unit: Participants] | 18
Current RLS medications, n (%) - Oxycodone [Count of Participants; unit: Participants] | 2
Current RLS medications, n (%) - Dopamine agonist [Count of Participants; unit: Participants] | 4
Current RLS medications, n (%) - Alpha-2-delta ligand [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Without a Clinically Significant Increase in RLS Symptoms During the First Phase Involving an Opioid Dose Reduction of >= 20% Relative to Baseline.
Description: Percentage of subjects without a clinically significant increase in RLS symptoms during the first Phase involving an opioid dose reduction of >= 20% relative to baseline. The clinically significant increase was assessed by determining the Clinician Global Impression of Improvement (CGI-I) score for the subject. Possible choices (followed by scale value) are: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very Much Worse (7). Scores of 6 or 7 would be considered a clinically significant increase in RLS Symptoms.
Time Frame: Week 1
Population: All eligible subjects who passed screening and were enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
Participants | 14

2. Secondary Outcome: Percentage of Subjects Without a Clinically Significant Increase in RLS Symptoms During the First Phase Involving an Opioid Dose Reduction of >= 1/3 Relative to Baseline.
Description: Percentage of subjects without a clinically significant increase in RLS symptoms during the first Phase involving an opioid dose reduction of >= 1/3 relative to baseline. The clinically significant increase was assessed by determining the Clinician Global Impression of Improvement (CGI-I) score for the subject. Possible choices (followed by scale value) are: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very Much Worse (7). Scores of 6 or 7 would be considered a clinically significant increase in RLS Symptoms.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 14
Participants | 8

3. Secondary Outcome: Change From Baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score During Step-down #1 With an Opioid Dose Reduction of >=20%
Description: IRLS is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe.
Time Frame: 1 week
Population: These 19 subjects entered step-down #1, but 1 of the original 20 reduced their medication by 17% and so was not included in the analysis population for this secondary outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 19
units on a scale | 5.8 (6.1)

4. Secondary Outcome: Change From Baseline in International Restless Legs Syndrome Study Group Rating Scale (IRLS) Score During Step-down #2 With an Opioid Dose Reduction of >=1/3
Description: IRLS is a participant-rated questionnaire that rates RLS severity from 0-40, where 40 is the most severe.
Time Frame: 1 week into Step-down #2
Population: The analysis population for this endpoint did not include the 3 subjects who were instructed to reduce opioid dose by >= 1/3 but actually reduced opioid dose by < 1/3 nor the 3 subjects who never were instructed to reduced opioid dose by >= 1/3 due to dropout before that phase. Data were missing from one subject and Last Observation Carried Forward (LOCF) was used for imputation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 14
units on a scale | 5.7 (6.9)

5. Secondary Outcome: Maximum Percent Change in Opioid Dose Relative to Baseline Without a Clinically Significant Increase in RLS Symptoms.
Description: The clinically significant increase was assessed by determining the Clinician Global Impression of Improvement (CGI-I) score for the subject. Possible choices (followed by scale value) are: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very Much Worse (7). Scores of 6 or 7 would be considered a clinically significant increase in RLS Symptoms.
Time Frame: 1 week into final step-down
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
percent change | 29.9 (23.7)

6. Other Pre Specified Outcome: NPNS Tolerability Rate - Percentage of Subjects Who Withdrew From Optional Phase 3 Citing Lack of Tolerability of NPNS as the Primary Reason for Withdrawal.
Description: Percentage of subjects who withdraw from study prior to the optional Phase 3 citing lack of tolerability of NPNS as the primary reason for withdrawal. The criterion for success was fewer than 20% of subjects who begin NPNS treatment withdrawing for this reason.
Time Frame: Up to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
Participants | 0

7. Other Pre Specified Outcome: Percentage of Grade 2 or Higher NPNS-related Adverse Events.
Description: A Grade 2 adverse event is described as: moderate; minimal, local, or non-invasive intervention indicated; limiting age appropriate instrumental Activities of Daily Living such as preparing meals, shopping for groceries or clothes, using the telephone, and managing money. The success criteria was fewer than 20% Grade 2 or higher NPNS-related adverse events. (Definition from the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 NCI, NIH, US Department of Health and Human Services (DHHS). May 29, 2009 NIH publication #- 09-7473.)
Time Frame: Up to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
Participants | 0

8. Other Pre Specified Outcome: Percentage of Grade 3 or Higher NPNS-related Adverse Events.
Description: The criteria for success were no Grade 3 or higher NPNS-related adverse events. A Grade 3 adverse event was described as: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care Activities of Daily Living such as bathing, dressing and undressing, feeding oneself, using the toilet, taking medications, and not being bedridden. (Definition from the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 NCI, NIH, DHHS. May 29, 2009 NIH publication #- 09-7473.)
Time Frame: Up to 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 20
Participants | 0

9. Other Pre Specified Outcome: NPNS Adherence Ratio During Step-down #1 and Step-down #2.
Description: NPNS adherence was based on the percent of device usage on nights with RLS symptoms during Assessment periods. Adherence was assessed during assessment periods based on objective electronic records of completed device sessions. Subjects were instructed to complete a device session on all days with RLS symptoms. The global criterion for success percentage was >=70%. The adherence ratio is the average days per week subjects completed device sessions divided by the average number of days that subjects experienced RLS symptoms.
Time Frame: 1 week post step-down
Measure: Mean (Standard Deviation); unit: percentage of days per week with RLS
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
Number analyzed (Participants) | 14
percentage of days per week with RLS | 85 (24)

ADVERSE EVENTS:
Time Frame: Up to 9 weeks
Arm/Group | Noninvasive Peripheral Nerve Stimulation (NPNS)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Noninvasive Peripheral Nerve Stimulation (NPNS) (N=20)
Discomfort (General disorders) | 9 (9)
Restless Legs Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) — Increased RLS symptoms due to Reduction in medication.
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT04698343/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04698343/ICF_001.pdf